CLINICAL TRIAL: NCT01336387
Title: A Randomized, Double-Blind, Single-dose and Multi-dose Study of the Novel Retinoid, 9cUAB30, to Determine Pharmacokinetics and Safety
Brief Title: Dose-Finding of Retinoid 9cUAB30 in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCI-2013-00468; CO10311; N01CN35153 (NIH)
Record Dates: First submitted 2011-03-24; First posted 2011-04-15 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2013-05

CONDITIONS: Healthy, no Evidence of Disease
MeSH Terms: interventions — UAB 30

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Arm I (retinoid 9cUAB30) (Experimental): Participants receive retinoid 9cUAB30* PO on days 1-28.
  Interventions: Drug: retinoid 9cUAB30; Other: pharmacological study; Other: laboratory biomarker analysis; Other: cancer prevention
- Arm II (placebo) (Placebo Comparator): Participants receive placebo* PO on days 1-28.
  Interventions: Other: placebo; Other: pharmacological study; Other: laboratory biomarker analysis; Other: cancer prevention

INTERVENTIONS:
Drug: retinoid 9cUAB30 — Given PO
  Arms: Arm I (retinoid 9cUAB30)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies
Other: cancer prevention — Disease prevention
  Other Names: cancer prevention intervention

SUMMARY:
This randomized phase I trial studies the side effects and the best dose of retinoid 9cUAB30 in healthy volunteers. Chemoprevention is the use of certain drugs to keep cancer from forming. The use of retinoid 9cUAB30 may keep cancer from forming.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary objective is to determine the toxicities and recommended phase II dose of 9cUAB30. The co- primary objective is to characterize the urine and plasma single dose and steady state pharmacokinetics of 9cUAB30 in normal volunteers.

SECONDARY OBJECTIVES:

I. To correlate the pharmacokinetics of 9cUAB30 with toxicity. II. To compare observed toxicity between placebo controls and each dose level. III. To assess for any change in single dose PK after repeat dosing (Day 1 vs. Day 36).

IV. To assess the following potential biomarkers of UAB30:

* Telomerase activity (measurement of telomeric repeats) in PBMCs.
* Gene expression of DNA methyltransferase in PBMCs.
* Gene expression of CYP2B6 in PBMCs.

OUTLINE: This is a dose-escalation study. Participants are randomized to 1 of 2 treatment arms.

ARM I: Participants receive retinoid 9cUAB30* orally (PO) on days 1-28.

ARM II: Participants receive placebo* PO on days 1-28.

Courses repeat every 28 days in the absence of unacceptable toxicity.

*NOTE: Participants receive doses on days 8, 15, 22 and 29 after they have fasted for 12 hours.

After completion of study treatment, patients are followed up on days 7 and 30.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status =< 1 (Karnofsky >= 70%)
* WBC >= 3000/mm^3
* Platelets >= 100,000mm^3
* Bilirubin =< upper limit of institutional normal
* AST =< upper limit of institutional normal
* Creatinine within institutional normal limits
* Sodium =< upper limit of institutional normal
* Potassium =< upper limit of institutional normal
* Chloride =< upper limit of institutional normal
* Bicarbonate =< upper limit of institutional normal
* Fasting triglycerides =<1.5 x ULN
* Fasting cholesterol =< 1.5 x ULN
* Participants must agree to discontinue all vitamin supplements while taking study medication and for thirty days past the last dose of study medication
* The effects of 9cUAB30 on the developing human fetus are unknown; for this reason, women must agree to use TWO effective forms of birth control for the duration of study participation and for 30 days following the last dose of study medication

  * The following persons are not considered to be able to father or bear children and therefore are eligible to participate without the use of concurrent birth control:

    * Female with bilateral oophorectomy and/or hysterectomy
    * Female with fallopian tubes cut, tied, or sealed
    * Female with sterilization implant (e.g. Adiana, Essure) placed > 3 months prior to randomization
    * Female post-menopausal (> 1 year since last menses)
    * Male with vasectomy > 3 months prior to randomization
  * One of the following methods of birth control must be used by women of childbearing potential:

    * Combined oral contraceptive pill in continuous use for > 30 days prior to study entry
    * Vaginal ring (e.g. NuvaRing) in continuous use for > 30 days prior to study entry
    * Skin patch (e.g. Ortho Evra) in continuous use for > 30 days prior to study entry
    * Injection (e.g. Depo-Provera, Noristerat®) in continuous use for > 30 days prior to study entry
    * Copper IUD (e.g. ParaGard)
  * Note: because of the decreased effectiveness of low dose progesterone-only contraceptive methods when used with retinoids, the following hormonal methods are NOT acceptable:

    * Low dose progesterone only oral contraceptive pill ("mini pills" e.g. Micronor®, Nor-Q.D., Ovrette)
    * Norplant subdermal implant
    * Mirena® Hormonal Implanted Uterine Device (IUD)
  * In addition to the above method of contraception, one of the following methods of contraception will ALSO be used for the duration of study participation and for 30 days following the last dose of study medication:

    * Diaphragm, cervical cap, or cervical shield with spermicide
    * Contraceptive sponge (e.g. Today Sponge)
    * Condom (male or female type) plus spermicide
* Females of child-bearing potential must have a negative pregnancy test within the current menstrual cycle and within 7 days before starting drug
* Participants must have the ability to understand, and the willingness to sign, a written informed consent document

Exclusion Criteria:

* Participants may not be taking medications that might interact with 9cUAB30; detailed list of potentially interacting medications
* Participants may not be taking lipid lowering agents
* Participants may not be receiving any other investigational agents
* Participants with a history of allergic reactions attributed to compounds of similar chemical or biologic composition of retinoids
* Participants with an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with 9cUAB30, breastfeeding must be discontinued for the duration of study participation and for one month after the last dose of the study agent if the mother is treated with 9cUAB30
* Individuals known to be HIV-positive may not participate in this study; the uncertain immune status of HIV-positive people and the potential risks of taking part in this study are too great to justify this non-treatment therapy
* Individuals with a history of cancer diagnosis or reoccurrence < 5 years from study entry may not participate; however, individuals with a history of squamous or basal cell carcinoma of the skin < 5 years from study entry will not be excluded from this study; the effects of this study agent on the immune system of people at risk for recurring cancer are unknown

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose of 9cUAB30 based on the MTD | 28 days
Pharmacokinetics of 9cUAB30 in normal volunteers | Baseline, days 1, 8, 15, 22, 36, and 43
  Using one-sample t-tests, or Wilcoxon signed-rank tests as appropriate in order to evaluate the single vs. steady state levels. An appropriate regression model will be used to explore the relationship of dose with change in PK.

SECONDARY OUTCOMES:
Correlation between pharmacokinetic and toxicity as assessed by CTCAE | Up to 36 days
Comparison of toxicity between placebo and controls as assessed by CTCAE | Up to 36 days
  To compare toxicities at each dose level to placebo, the Chi-square test will be used for the presence or absence of toxicities, and Wilcoxon rank-sum tests will be used for CTCAE grade and investigator defined relationship data.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Kolesar, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States